CLINICAL TRIAL: NCT01431950
Title: A Randomised, Double-blind, Multi-centre Study to Evaluate the Efficacy and Safety of Inhaled Fluticasone Furoate in the Treatment of Persistent Asthma in Adults and Adolescents Currently Receiving Mid to High Strength Inhaled Corticosteroids.
Brief Title: Evaluating the Efficacy and Safety of Fluticasone Furoate in the Treatment of Asthma in Adults and Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 114496
Record Dates: First submitted 2011-08-25; First posted 2011-09-12 (Estimated); Results first posted 2014-09-03 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
Keywords: fluticasone furoate
MeSH Terms: conditions — Asthma | interventions — fluticasone furoate; Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FF 100mcg once daily (Experimental): Inhaled corticosteroid (ICS)
  Interventions: Drug: fluticasone furoate; Drug: albuterol/salbutamol
- FF 200mcg once daily (Experimental): Inhaled corticosteroid
  Interventions: Drug: fluticasone furoate; Drug: albuterol/salbutamol

INTERVENTIONS:
Drug: fluticasone furoate — Inhaled corticosteroid
Drug: albuterol/salbutamol — Provided as rescue relief of asthma symptoms

SUMMARY:
A randomised, double-blind, multi-centre study to evaluate the efficacy and safety of two doses of inhaled fluticasone furoate in the treatment of persistent asthma in adults and adolescents currently receiving mid to high strength inhaled corticosteroids.

DETAILED DESCRIPTION:
This will be a multi-centre, randomised, double-blind, parallel-group study. Subjects meeting all the inclusion criteria and none of the exclusion criteria during Visit 1 (screening visit) will enter a four week Run-In period during which they will remain on their baseline ICS medication. In addition, all subjects will be provided with albuterol/salbutamol for relief of asthma symptoms. Subjects failing screening will not be eligible for re-screening. During the Run-In and double-blind treatment periods subjects will maintain an electronic daily diary to record morning and evening Peak Expiratory Flow (PEF), asthma symptom score and rescue albuterol/salbutamol use. Subjects will receive a contact (Phone Contact 1/optional office visit (1b)) during Run-In to reinforce compliance with Run-In medication and diary monitoring. Those subjects who meet the eligibility criteria at the end of the Run-In period will be stratified in an approximately 1:1 ratio according to their baseline FEV1 as a percentage of predicted normal - one stratum for those with FEV1 percent predicted ≥40% to ≤65% and one for those with FEV1 percent predicted >65% to ≤90%. Once stratified, subjects will be randomised to one of the following treatments and enter into a 24 week double-blind treatment period:1) Fluticasone furoate 100mcg once daily in the evening or 2) Fluticasone furoate 200mcg once daily in the evening.

Subjects will then attend 6 on-treatment visits at Visits 3, 4, 5, 6, 7 and 8 (Weeks 2, 4, 8, 12, 18 and 24 respectively). All visits including Visit 1 must be conducted in the evening between 5 PM and 11 PM. Subjects will receive treatment for 24 weeks. Twenty four hour urinary cortisol assessments will be collected at the end of Run-In (Visit 2) and at end of treatment (Visit 8) visits. A follow-up contact will be performed 1-week after completing study medication (Visit 9). Subjects will participate in the study for up to a maximum of 29 weeks (including screening, treatment and follow-up contact). In addition, partially used NDPIs will be collected in a subset of subjects. For subjects who have consented for pharmacogenetics, a blood sample will also be taken for pharmacogenetic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Outpatient at least 12 years of age with diagnosis of asthma at least 12 weeks prior to first visit
* Both genders; females of child bearing potential must be willing to use appropriate contraception
* Pre-bronchodilator FEV1 of 40-90% predicted
* Reversibility FEV1 of at least 12% and 200mLs
* Current asthma therapy that includes inhaled corticosteroid for at least 4 weeks prior to first visit

Exclusion Criteria:

* History of life threatening asthma
* Respiratory infection or candidiasis
* Asthma exacerbation requiring OCS within last 4 weeks or overnight hospital stay within the last 3 months
* Concurrent respiratory disease or other disease that would confound study participation of affect subject safety
* Allergies to study drugs, study drug excipients, medications related to study drugs
* Taking another investigational medication or medication prohibited for use during the study
* Previous treatment with FF or FF/VI in a phase II or III study
* Night shift workers
* Children in care

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2011-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (38):
- United States (19):
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Albany, Georgia
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, Bethesda, Maryland
  - GSK Investigational Site, Plymouth, Minnesota
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Brick, New Jersey
  - GSK Investigational Site, Utica, New York
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Corsicana, Texas
- Argentina (3):
  - GSK Investigational Site, Mendoza, Mendoza Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, San Miguel de Tucumán
- Chile (3):
  - GSK Investigational Site, Valparaíso, Región de Valparaíso
  - GSK Investigational Site, Puente Alto - Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago, Región Metro de Santiago
- France (6):
  - GSK Investigational Site, Aigrefeuille-sur-Maine
  - GSK Investigational Site, Bourg-des-Comptes
  - GSK Investigational Site, Châlons-en-Champagne
  - GSK Investigational Site, Laon
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Vannes
- Mexico (2):
  - GSK Investigational Site, Villahermosa, Tabasco
  - GSK Investigational Site, Mexico City
- Russia (5):
  - GSK Investigational Site, Belgorod
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Novokuznetsk
  - GSK Investigational Site, Penza
  - GSK Investigational Site, Pyatigorsk

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] O'Byrne PM, Jacques L, Goldfrad C, Kwon N, Perrio M, Yates LJ, Busse WW. Integrated safety and efficacy analysis of once-daily fluticasone furoate for the treatment of asthma. Respir Res. 2016 Nov 24;17(1):157. doi: 10.1186/s12931-016-0473-x. PMID 27881132
- [Derived] Woodcock A, Lotvall J, Busse WW, Bateman ED, Stone S, Ellsworth A, Jacques L. Efficacy and safety of fluticasone furoate 100 mug and 200 mug once daily in the treatment of moderate-severe asthma in adults and adolescents: a 24-week randomised study. BMC Pulm Med. 2014 Jul 9;14:113. doi: 10.1186/1471-2466-14-113. PMID 25007865
- [Derived] Svedsater H, Jacques L, Goldfrad C, Bleecker ER. Ease of use of the ELLIPTA dry powder inhaler: data from three randomised controlled trials in patients with asthma. NPJ Prim Care Respir Med. 2014 Jun 26;24:14019. doi: 10.1038/npjpcrm.2014.19. No abstract available. PMID 24966061
- [Derived] Svedsater H, Dale P, Garrill K, Walker R, Woepse MW. Qualitative assessment of attributes and ease of use of the ELLIPTA dry powder inhaler for delivery of maintenance therapy for asthma and COPD. BMC Pulm Med. 2013 Dec 7;13:72. doi: 10.1186/1471-2466-13-72. PMID 24314123
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 114496 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114496 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114496 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114496 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114496 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114496 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114496 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants meeting eligibility criteria at the Screening visit entered a 4-week Run-in Period for Baseline safety evaluations and to obtain measures of asthma status. Participants were then randomized to a 24-week Treatment Period. A total of 500 participants were screened; 239 were randomized, and 238 received >=1 dose of study treatment.
Groups:
- FF 100 µg OD: Participants received fluticasone furoate (FF) 100 micrograms (µg) inhalation powder via a Dry Powder Inhaler (DPI) once daily (OD) in the evening for 24 weeks. In addition, all participants were provided with albuterol/salbutamol aerosol to be used as rescue medication as needed.
- FF 200 µg OD: Participants received FF 200 µg via a DPI OD in the evening for 24 weeks. In addition, all participants were provided with albuterol/salbutamol aerosol to be used as rescue medication as needed.
Period: Overall Study
Arm/Group | FF 100 µg OD | FF 200 µg OD
Started | 119 | 119
Completed | 100 | 104
Not Completed | 19 | 15
Not completed — Study Site Closed/Terminated | 7 | 3
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Protocol Violation | 2 | 3
Not completed — Adverse Event | 2 | 2
Not completed — Physician Decision | 2 | 1
Not completed — Lack of Efficacy | 2 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Met Protocol-defined Stopping Criteria | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FF 100 µg OD | FF 200 µg OD | Total
Number analyzed (Participants) | 119 | 119 | 238
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.6 (15.41) | 45.1 (15.78) | 45.9 (15.58)
Gender [Count of Participants; unit: Participants]
  Female | 81 | 79 | 160
  Male | 38 | 40 | 78
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage (HER) | 5 | 4 | 9
  Central/South Asian HER | 1 | 0 | 1
  Japanese/East Asian HER /South East Asian HER | 0 | 3 | 3
  Native Hawaiian or other Pacific Islander | 1 | 0 | 1
  White | 101 | 100 | 201
  American Indian or Alaska Native & White | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Clinic Visit Evening (Pre-bronchodilator and Pre-dose) Forced Expiratory Volume in One Second (FEV1) at the End of the 24-week Treatment Period
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Evening clinic visit FEV1 is defined as the clinic visit (pre-bronchodilator and pre-dose) FEV1 measurement taken at the Week 24 clinic visit. Pre-dose and pre-rescue albuterol/salbutamol trough FEV1 were measured electronically by spirometry in the evening at the Baseline through Week 24 clinic visits. The highest of 3 technically acceptable measurements was recorded. Baseline was the pre-dose value obtained at Visit 2. Change from Baseline was calculated as the Week 24 value minus the Baseline value. Analysis was performed using analysis of covariance (ANCOVA) with covariates of Baseline, region, sex, age, and treatment. The last observation carried forward (LOCF) method was used to impute missing data, in which the last non-missing, pre-dose, post-Baseline on-treatment measurement at scheduled clinic visits was used to impute the missing value.
Time Frame: Baseline and Week 24
Population: Intent-to-Treat (ITT) Population: all participants (par.) randomized to treatment who received >=1 dose of study medication, except for the par. of one investigator (excluded after good clinical practice [GCP] issues identified during a site audit). Only those par. with non-missing covariates and post-Baseline FEV1 data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | FF 100 µg OD | FF 200 µg OD
Number analyzed (Participants) | 106 | 109
Liters | 0.208 (0.0417) | 0.284 (0.0411)
Statistical Analysis 1: Comparison: FF 100 µg OD vs FF 200 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.077, 95% CI [-0.039 to 0.192]

2. Secondary Outcome: Change From Baseline in the Percentage of Rescue-free 24-hour (hr) Periods Over the 24-week Treatment Period
Description: The number of inhalations of rescue bronchodilator, albuterol/salbutamol inhalation aerosol, used during the day and night was recorded by the participants in a daily electronic diary (eDiary). A 24-hour period in which a participant's responses to both the morning and evening assessments indicated no use of rescue medication was considered to be rescue free. A 24-hour period was considered as missing if both day time and night time values were missing or if one of the day time or night time values were missing and the other value indicated no use of rescue medication. The Baseline value is the average of the values over the last 7 days of the daily eDiary prior to the randomization of the participant. Change from Baseline was calculated as the averaged value during the 24-week Treatment Period minus the Baseline value. Analysis was performed using ANCOVA with covariates of Baseline, region, sex, age, and treatment.
Time Frame: From Baseline up to Week 24
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of rescue-free 24-hr periods
Arm/Group | FF 100 µg OD | FF 200 µg OD
Number analyzed (Participants) | 108 | 109
Percentage of rescue-free 24-hr periods | 21.3 (3.05) | 23.1 (3.03)

3. Secondary Outcome: Change From Baseline in Daily Evening (PM) Peak Expiratory Flow (PEF) Averaged Over the 24-week Treatment Period
Description: PEF is a measure of lung function and is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. PEF was measured by the participants using a hand-held electronic peak flow meter each morning and evening prior to the dose of study medication and any rescue albuterol/salbutamol inhalation aerosol use. Change from Baseline (defined as the average of the values of the last 7 days prior to randomization of the participants) was calculated as the value of the averaged daily trough PM PEF over the 24-week Treatment Period minus the Baseline value. Analysis was performed using ANCOVA with covariates of Baseline, region, sex, age, and treatment.
Time Frame: From Baseline up to Week 24
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters/minute (L/min)
Arm/Group | FF 100 µg OD | FF 200 µg OD
Number analyzed (Participants) | 108 | 109
Liters/minute (L/min) | 5.9 (3.26) | 7.2 (3.25)

4. Secondary Outcome: Change From Baseline in Daily Morning (AM) PEF Averaged Over the 24-week Treatment Period
Description: PEF is a measure of lung function and is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. PEF was measured by the participants using a hand-held electronic peak flow meter each morning and evening prior to the dose of study medication and any rescue albuterol/salbutamol inhalation aerosol use. Change from Baseline (defined as the average of the values of the last 7 days prior to randomization of the participants) was calculated as the value of the averaged daily AM PEF over the 24-week Treatment Period minus the Baseline value. Analysis was performed using ANCOVA with covariates of Baseline, region, sex, age, and treatment.
Time Frame: From Baseline up to Week 24
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | FF 100 µg OD | FF 200 µg OD
Number analyzed (Participants) | 108 | 109
L/min | 13.4 (3.22) | 13.2 (3.20)

5. Secondary Outcome: Change From Baseline in the Percentage of Symptom-free 24-hour (hr) Periods Over the 24-week Treatment Period
Description: Asthma symptoms were recorded in a daily eDairy by the participants every day in the morning and evening before taking any rescue or study medication and before the peak expiratory flow measurement. A 24-hour period in which a participant's responses to both the morning and evening assessments indicated no symptoms was considered to be symptom free. A 24-hour period was considered as missing if both the day time and night time data were missing or if one was symptom-free but the other was missing. The Baseline value was the average of the values of the last 7 days of the daily eDiary prior to the randomization of the participant. Change from Baseline was calculated as the averaged value during the 24-week Treatment Period minus the Baseline value. Analysis was performed using ANCOVA with covariates of Baseline, region, sex, age, and treatment.
Time Frame: From Baseline up to Week 24
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of symptom-free 24-hr periods
Arm/Group | FF 100 µg OD | FF 200 µg OD
Number analyzed (Participants) | 108 | 109
Percentage of symptom-free 24-hr periods | 17.5 (2.80) | 19.6 (2.79)

ADVERSE EVENTS:
Time Frame: On-treatment adverse events (AEs), defined as those events occurring while participants were on treatment, up to and including the day after the last dose (up to 24 weeks), are reported.
Description: Serious AEs (SAEs) and non-serious AEs were collected in the Safety Population, comprised of all participants randomized to treatment who received at least one dose of study medication.
Arm/Group | FF 100 µg OD | FF 200 µg OD
Serious Adverse Events (participants affected / at risk) | 3/119 | 4/119
Other Adverse Events (participants affected / at risk) | 52/119 | 49/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FF 100 µg OD (N=119) | FF 200 µg OD (N=119)
Chondromalacia (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1
Abscess (Infections and infestations) | 0 | 1
Acute sinusitis (Infections and infestations) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FF 100 µg OD (N=119) | FF 200 µg OD (N=119)
Nasopharyngitis (Infections and infestations) | 14 | 15
Bronchitis (Infections and infestations) | 14 | 8
Influenza (Infections and infestations) | 5 | 8
Sinusitis (Infections and infestations) | 8 | 5
Pharyngitis (Infections and infestations) | 7 | 4
Upper respiratory tract infection (Infections and infestations) | 2 | 7
Headache (Nervous system disorders) | 12 | 15
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.